CLINICAL TRIAL: NCT04126967
Title: Next Generation Sequencing（NGS）Monitors Minimal Residual Disease（MRD）in Allo-PBSCT Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xianmin Song, MD (Other)
Responsible Party: Sponsor-Investigator, Xianmin Song, MD, chief of hematology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHSYXY- NGS-2019003
Record Dates: First submitted 2019-10-07; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: NGS Monitor MRD
Keywords: NGS; MRD; Allo-PBSCT

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allo-PBSCT patients with no NGS text (Other)
  Interventions: Diagnostic Test: NGS patients

INTERVENTIONS:
Diagnostic Test: NGS patients — The next generation sequencing technique (NGS) was used to monitor the minimal residual lesions after allogeneic hematopoietic stem cell transplantation

SUMMARY:
Objective: to evaluate the value of high-throughput next generation gene sequencing (NGS) in the detection of minimal residual disease (MRD) and recurrence after allogeneic transplantation.

Overview of study design. This study is a single-center, single-arm, prospective clinical trial designed to evaluate the significance of next generation gene sequencing (NGS) in monitoring for minimal residual disease (MRD) and recurrence after allogeneic transplantation.

This clinical study is observational and does not involve drugs. Next generation sequencing (NGS) were used to monitor minor residual lesions after allogeneic hematopoietic stem cell transplantation, to predict disease recurrence early, and to monitor and evaluate prognosis, so as to provide basis for early intervention treatment after transplantation, so as to reduce hematological recurrence and improve survival rate.

This clinical study is observational and does not involve drugs.The sensitive next generation sequencing (NGS) was used to monitor the minimal residual lesions after allogeneic hematopoietic stem cell transplantation, to predict the relapse of the disease in the early stage, and to monitor and evaluate the prognosis, so as to provide the basis for early intervention treatment after transplantation, so as to reduce the hematological relapse and improve the survival rate.

DETAILED DESCRIPTION:
Minimal residual disease (MRD) detection is the detection of residual micro-clones in patients with leukemia in remission, predicting the recurrence of the disease, and determining the next treatment of the disease.There are many methods to detect MRD, the most common one is Flow cytometry (FCM).The fusion genes of Wilms tumor 1（WT1）, pml-rara, runx1-runx1t1, cbfb-myh11 and nucleophosmin(NPM1) were detected by Polymerase Chain Reaction(PCR).Chromosome analysis;Fluorescence in situ hybridization（FISH）, etc.FCM is a commonly used method for clinical detection of MRD, with a sensitivity of 10-3~ 4. Its specificity is only high when there is abnormal cloning in specimens, and false negative can be caused when there is phenotypic drift and bone marrow dilution.PCR detection of WT1 is considered to be a marker of preleukaemia, but WT1 is also expressed in non-leukemic cells and is not recommended by the European leukaemia network (ELN).PCR detection of pml-rara, runx1-runx1t1, cbfb-myh11 and other fused genes only supported the clinical trial data when the log index decreased in the numerical procedure.Chromosome analysis is less sensitive because of its lack of metaphase chromosome division.FISH has a sensitivity of 10-2~ 3, specificity is only high in abnormal cells, but detection rate of mutations not covered by probes is low, and non-specific binding of probes can lead to false positives.The sensitivity, specificity and pertinence of various MRD detection technologies are different. Currently, these technologies are combined to analyze MRD clinically.

Next generation gene sequencing (NGS) is the ability to simultaneously detect the structure of all disease clones and subclones and track their changing mutations.Compared with PCR and FCM that detect abnormalities in a single clone, NGS can detect each disease clone and subclone.NGS has been clinically used to diagnose mutations and subtypes of blood diseases.Persistent mutations are associated with high recurrence rates.

This clinical study is observational and does not involve drugs.The sensitive next generation sequencing (NGS) was used to monitor the minimal residual lesions after allogeneic hematopoietic stem cell transplantation, to predict the relapse of the disease in the early stage, and to monitor and evaluate the prognosis, so as to provide the basis for early intervention treatment after transplantation, so as to reduce the hematological relapse and improve the survival rate.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, male or female;
2. Patients who received allogeneic peripheral blood hematopoietic stem cell transplantation ;
3. Patients must be able to understand and be willing to participate in this study and sign informed consent.-

Exclusion Criteria:

1. Non-allogeneic hematopoietic stem cell transplantation patients;
2. The expected survival rate is less than 3 months after transplantation;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
NGS results | 3 years
  positive: VAF>0.2%; negative: VAF <0.1%
MRD by FCM | 3 years
  posotive：MRD by FCM≥0.01%， negative:MRD by FCM<0.01%
Donor chimerism (DC) | 3 years
  positive: the chimerism rate increased ((STR < 90%) or FISH > 0.6%);negative:chimerism rate reached(STR > 95% or xy-FISH Donor chromosome > 99.4%)
fusion gene or WT1 | 3 years
  positive:WT1/ reference gene, bone marrow >2%;negative:negative fusion gene, WT1/ reference gene <0.6%.
relapse | 3 years
  The number of patients relapse after Allo-PBSCT

SECONDARY OUTCOMES:
survival | 3 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China